CLINICAL TRIAL: NCT03296176
Title: Metabolomic Study in Huntington's Disease
Brief Title: Metabolomic Study in Huntington's Disease (METABO-HD)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 49RC17_0086
Record Dates: First submitted 2017-09-15; First posted 2017-09-28 (Actual); Last update posted 2017-11-01 (Actual); Status verified 2017-09

CONDITIONS: Huntington Disease
MeSH Terms: conditions — Huntington Disease | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- presymptomatic (Experimental)
  Interventions: Biological: blood sample
- symptomatic (Experimental)
  Interventions: Biological: blood sample
- controls (Other)
  Interventions: Biological: blood sample

INTERVENTIONS:
Biological: blood sample — blood sample for metabolome analyse

SUMMARY:
The purpose of this project is to study Huntington's disease by metabolomic approach.

ELIGIBILITY:
Inclusion Criteria:

For all groups:

* age between 20 and 70 years
* signature of the informed consent
* covered by social security

For presymptomatic group:

* positive genetic test with CAG repeat length ≥ 37 in HTT gene
* Unified Huntington Disease Rating Scale ≤ 5

For symptomatic group:

* positive genetic test with CAG repeat length ≥ 37 in HTT gene
* The Unified Huntington's Disease Rating Scale motor score ≥ 6
* The Total Functional Capacity score ≥ 11

Exclusion Criteria for all groups:

* participation in another therapeutic trial (3 months exclusion period)
* pregnancy and breastfeeding
* persons deprived of their liberty by judicial or administrative decision

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2017-10-09 (Actual); Primary Completion 2019-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
metabolite mass | at baseline
  by chromatography and mass spectrometry

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Verny, PU-PH, Principal Investigator — University Hospital, Angers
Locations (1):
- CHU Angers, Angers, France